CLINICAL TRIAL: NCT01604395
Title: An Open, Multi-center, Prospective and Retrospective Observational Study to Evaluate the Long-term Safety and Effectiveness of Growth Hormone (Eutropin Inj. / Eutropin Plus Inj.) Treatment With GHD, TS, CRF, SGA, ISS and PWS in Children
Brief Title: Long-term Safety and Effectiveness of Growth Hormone With GHD, TS, CRF, SGA , ISS and PWS in Children
Acronym: LGS
Status: Recruiting | Type: Observational
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Other Study IDs: LG-HGOS001
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Growth Hormone Deficiency; Turner Syndrome; Chronic Renal Failure; Small for Gestational Age; Idiopathic Short Stature
Keywords: GHD; TS; CRF; SGA; ISS; PWS
MeSH Terms: conditions — Dwarfism, Pituitary; Turner Syndrome; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- growth hormone

SUMMARY:
The purpose of this study is to evaluate the long-term safety and effectiveness of growth hormone (Eutropin Inj./Eutropin plus Inj.) treatment with GHD (Growth Hormone Deficiency), TS (Turner Syndrome),CRF (Chronic Renal Failure), SGA (Small for Gestational Age), and ISS (Idiopathic Short Stature).

ELIGIBILITY:
Inclusion Criteria:

* short stature children aged 2 years or more
* children with GHD,TS, CRF, SGA or ISS
* written informed consent from the person, person's parent or legal guardian

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children with GHD, TS, CRF, SGA and ISS
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2012-01; Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety measure : adverse event | up to 2 years after epiphyseal closure

SECONDARY OUTCOMES:
effectiveness measure : difference in target height and final height | up to 2 years after epiphyseal closure
effectiveness : difference in height velocity between Baseline and every year | up to 2 years after epiphyseal closure
effectiveness measure : difference in height SDS for CA between baseline and every 6 months | up to 2 years after epiphyseal closure

CONTACTS AND LOCATIONS:
Overall Officials: HW Chae, M.D., Principal Investigator — Kangnam severance hospital; KS Sim, M.D., Principal Investigator — Kangdong KyungHee University hospital; IT Hwang, M.D., Principal Investigator — Kangdong Sacred Heart Hospital; SC Chung, M.D., Principal Investigator — Konkook University hospital; CW Ko, M.D., Principal Investigator — Kyungpook National University Hospital; HS Kim, M.D., Principal Investigator — Keimyung University hospital; YJ Lee, M.D., Principal Investigator — Korea University; KH Lee, M.D., Principal Investigator — Korea University Anam Hospital; JH Lee, M.D., Principal Investigator — Kosin university hospital; JS Yu, M.D., Principal Investigator — Dankook University; JH Yu, M.D., Principal Investigator — Dong-A University Hospital; SY Lee, M.D., Principal Investigator — SMG-SNU Boramae Medical Center; WY Chung, M.D., Principal Investigator — Inje University; Yl Shin, M.D., Principal Investigator — Buchun Soonchunhyang university hospital; CY Kim, M.D., Principal Investigator — daejin medical center; DK Jin, M.D., Principal Investigator — Samsung Medical Center; MJ Park, M.D., Principal Investigator — Inje University; CH Shin, M.D., Study Chair — Seoul National University Hospital; BK Suh, M.D., Principal Investigator — Seoul St. Mary's Hospital; HW Yoo, M.D., Principal Investigator — Asan Medical Center; MH Jung, M.D., Principal Investigator — Yeouide St. Mary's hospital; SH Park, M.D., Principal Investigator — St Vincent's Hospital; DH Kim, M.D., Principal Investigator — Sowha children's hospital; DH Lee, M.D., Principal Investigator — Seoul Soonchunhyang university hospital; HS Kim, M.D., Principal Investigator — Sinchon severance hospital; JS Hwang, M.D., Principal Investigator — Ajou University School of Medicine; SY Kim, M.D., Principal Investigator — Pusan National University Yangsan Hospital; JD Kim, M.D., Principal Investigator — Wonkwang university school of medicine & hospital; HS Han, M.D., Principal Investigator — Chungbuk National University Hospital; KH Lee, M.D., Principal Investigator — Wonkwang University Sanbon Medical Center; EK Yoo, M.D., Principal Investigator — Bunsangcha hospital; BK Lim, M.D., Principal Investigator — Wonju Christian Hospital; JH Kang, M.D., Principal Investigator — Eulji University Hospital; JY Seo, M.D., Principal Investigator — Eulji General Hospital; HS Kim, M.D., Principal Investigator — ehwa university medical center; JE Lee, M.D., Principal Investigator — Inha University Hospital; JH Kim, M.D., Principal Investigator — Inje University; CJ Kim, M.D., Principal Investigator — Chonnam National University Hospital; DY Lee, M.D., Principal Investigator — Chonbuk National University Hospital; KS Shin, M.D., Principal Investigator — Jeju National University Hospital; IT Hwang, M.D., Principal Investigator — Hallym University Medical Center; SM Lee, M.D., Principal Investigator — Hanyang University; KH Lee, M.D., Principal Investigator — Korea University Guro Hospital; KS Jo, M.D., Principal Investigator — Bucheon St. Mary's Hospital; SY Ahn, M.D., Principal Investigator — KangWon National University Hospital; PS Oh, M.D., Principal Investigator — Chuncheon Sacred Heart Hospital; S Yang, M.D., Principal Investigator — Hallym University Kangnam Sacred Heart Hospital; EY Kim, M.D., Principal Investigator — Chosun University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim JH, Kim SJ, Chung IH, Lim JS. Adiposity Rebound Timing in Small for Gestational Age Children Treated With Growth Hormone: Results From LG Growth Study Data. J Korean Med Sci. 2025 Feb 3;40(4):e12. doi: 10.3346/jkms.2025.40.e12. PMID 39901524
- [Derived] Jeong HR, Lee HS, Hwang JS. Growth Prediction Model for Prepubertal Children With Idiopathic Growth Hormone Deficiency: An Analysis of LG Growth Study Data. Clin Endocrinol (Oxf). 2025 Mar;102(3):281-287. doi: 10.1111/cen.15178. Epub 2024 Dec 15. PMID 39676465
- [Derived] Lee HS, Kum CD, Rho JG, Hwang JS. Long-term effectiveness of growth hormone therapy in children born small for gestational age: An analysis of LG growth study data. PLoS One. 2022 Apr 26;17(4):e0266329. doi: 10.1371/journal.pone.0266329. eCollection 2022. PMID 35472208
- [Derived] Lim HH, Kim YM, Lee GM, Yu J, Han HS, Yu J. Growth Responses During 3 Years of Growth Hormone Treatment in Children and Adolescents With Growth Hormone Deficiency: Comparison Between Idiopathic, Organic and Isolated Growth Hormone Deficiency, and Multiple Pituitary Hormone Deficiency. J Korean Med Sci. 2022 Mar 21;37(11):e90. doi: 10.3346/jkms.2022.37.e90. PMID 35315601
- [Derived] Cho WK, Ahn MB, Kim EY, Cho KS, Jung MH, Suh BK. Predicting First-Year Growth in Response to Growth Hormone Treatment in Prepubertal Korean Children with Idiopathic Growth Hormone Deficiency: Analysis of Data from the LG Growth Study Database. J Korean Med Sci. 2020 May 18;35(19):e151. doi: 10.3346/jkms.2020.35.e151. PMID 32419399